CLINICAL TRIAL: NCT03398239
Title: Dokuz Eylul University School of Medicine
Brief Title: Comparison of BPAP ST/T and BPAP ST / T Mode With AVAPS for Hypercapnic Respiratory Failure in ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Başak Bayram, Assistant Professor Dr., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2089357
Record Dates: First submitted 2016-11-30; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Hypercapnic Respiratory Failure
Keywords: respiratory failure, hypercapnia, BPAP, AVAPS
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BPAP ST/T (Active Comparator): Non-invasive Ventilation with BPAP ST/T mode
  Interventions: Device: Noninvasive mechanical ventilation
- AVAPS (Experimental): Non-invasive Ventilation with AVAPS mode
  Interventions: Device: Noninvasive mechanical ventilation

INTERVENTIONS:
Device: Noninvasive mechanical ventilation

SUMMARY:
The aim of the present study; To compare the effects of respiratory support options available for NIMV at the emergency department; i.e. AVAPS and ST/T modes, on the patient's pCO2 values, additional treatment need (another non-invasive ventilation method or endotracheal intubation) and the duration of stay in hospital.

DETAILED DESCRIPTION:
Non-invasive positive pressure ventilation (NIMV) is a life-saving procedure for patients with hypoxic and/or hypercapnic respiratory failure. AVAPS (average volume assured pressure support) is a noninvasive ventilation mode which has been developed to assure volume and pressure controlled respiratory support. AVAPS can ensure a constant tidal air volume to the patient with variable pressure support. Thus the positive features of the volume and pressure controlled support, which have a positive impact on the healing and recovery processes are combined.

This study aims to compare, in a randomized order, BPAP ST/T and BPAP ST / T Mode with AVAPS, in patients with hypercapnic respiratory failure in the emergency department.

Subjects: One hundred and two patients with hypercapnic respiratory failure will be included.

Primary outcome; decrease in the PaCO2 values

Secondary outcomes are stated as; Failure of treatment options, or change of the NIMV mode due to patient noncompliance or the patient's need for intubation and length of hospital stay (length of stay in the hospital from the emergency department).

ELIGIBILITY:
Inclusion Criteria:

PaCO2 > 45mmHg and any of the following

* SaO2 <90% on air
* SaO2 <93% on >6 Litres O2/min
* Inability to speak in sentences due to respiratory distress
* Respiratory rate > 24/min
* Altered mental status
* The use of accessory muscles of respiration

Exclusion Criteria:

* Respiratory arrest or unstable cardiorespiratory status
* Suspected Pneumothorax
* Urgent need for intubation
* Systolic blood pressure < 90 mmHg
* Inability to protect airway
* Facial deformity
* Facial, esophageal, or gastric surgery history
* All trauma patients
* Acute myocardial infarction
* Severe arrythmias
* Refractory nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
PaCO2 values | On arrival, at one hour, and at two hourly intervals thereafter
  Will measure change in PaCO2 values in the blood gase analysis of patients comparing those treated with BPAP ST/T and those with AVAPS

SECONDARY OUTCOMES:
Failure of treatment options | During the treatment
  Change of the NIMV mode due to patient noncompliance (switching to the second mode) or the patient's need for intubation during the treatment
Length of hospital stay | up to 6 months
  Length of hospital stay in the hospital (From the emergency department admission)
The time of treatment | During the treatment
  The sum of the noninvasive ventilation time in the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Bayram, MD, Study Director — Dokuz Eylul University, School of Medicine, Department of Emergency Medicine
Locations (1):
- Dokuz Eylul University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided